CLINICAL TRIAL: NCT06300255
Title: Evaluation of the H.O.O.V.E.S. Healing Intensives Program
Status: Recruiting | Type: Observational
Sponsor: VA Salt Lake City Health Care System (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: IRB 00166616
Record Dates: First submitted 2024-02-27; First posted 2024-03-08 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Anxiety; PTSD; Depression
Keywords: Horses; Anxiety; PTSD; Depression
MeSH Terms: conditions — Anxiety Disorders; Stress Disorders, Post-Traumatic; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- H.O.O.V.E.S. Healing Intensives Participants: Veterans enrolled in a H.O.O.V.E.S. healing intensives program and must have served in the military.
  Interventions: Behavioral: H.O.O.V.E.S. Healing Intensives

INTERVENTIONS:
Behavioral: H.O.O.V.E.S. Healing Intensives — "H.O.O.V.E.S. is a private, donor-supported charity dedicated to providing fully-funded, [4]-day, non-clinical healing intensives for veterans, their families and caregivers, and first responders across the nation who are seeking recovery from service-connected stress." 1
  References
  1. Home. HOOVES for Vets. Accessed January 24, 2024. https://www.hooves.us/.

SUMMARY:
The aim of this study is to measure the impact of these H.O.O.V.E.S. healing intensives on Veteran participants using several psychological instruments. The investigators are planning to administer the demographic questionnaires and psychological instruments to Veteran participants before the healing intensives. Psychological instruments will be administered immediately pre-intervention, pre- and post-session for each session, post-intervention, 90, 120 and 360 days post-intervention. The primary aim is to assess for statistically significant changes pre- to post session and pre- to post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* Veterans who have served in the military
* Must be enrolled in a H.O.O.V.E.S. Healing Intensives Program
* English speakers

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Veterans enrolled in a H.O.O.V.E.S. healing intensives program and must have served in the military.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2024-04-24 (Actual); Primary Completion 2029-02-01 (Estimated); Study Completion 2029-02-01 (Estimated)

PRIMARY OUTCOMES:
Mean Difference in AAQII pre- to post-session and pre- to post-intervention | through study completion, an average of 5 years
  AAQII is a 10-item measure that assesses psychological flexibility, with higher values indicating greater psychological inflexibility. The aim is to assess for statistically significant changes pre- to post session (1 day = a session) and pre- to post-intervention using paired t-test as well as ANCOVA adjusting for the significant demographic or diagnostic covariates.
Mean Difference in PANAS pre- to post-session and pre- to post-intervention | through study completion, an average of 5 years
  PANAS measures short-term positive and negative emotions. The aim is to assess for statistically significant changes pre- to post session (1 day = a session) and pre- to post-intervention using paired t-test as well as ANCOVA adjusting for the significant demographic or diagnostic covariates.
Mean Difference in STAI pre- to post-session and pre- to post-intervention | through study completion, an average of 5 years
  The STAI tracks the symptoms of anxiety, and the total score ranges from 20 to 80. The aim is to assess for statistically significant changes pre- to post session (1 day = a session) and pre- to post-intervention using paired t-test as well as ANCOVA adjusting for the significant demographic or diagnostic covariates.
Mean Difference in PCL pre- to post-session and pre- to post-intervention | through study completion, an average of 5 years
  PCL measures PTSD symptoms. The total PCL score can range from 17 to 85, with higher values indicating greater PTSD symptoms. The aim is to assess for statistically significant changes pre- to post session (1 day = a session) and pre- to post-intervention using paired t-test as well as ANCOVA adjusting for the significant demographic or diagnostic covariates.
Mean Difference in BDI pre- to post-session and pre- to post-intervention | through study completion, an average of 5 years
  The Beck Depression Inventory (BDI) measures depressive symptoms, with higher values indicating greater depressive symptoms. The aim is to assess for statistically significant changes pre- to post session (1 day = a session) and pre- to post-intervention using paired t-test as well as ANCOVA adjusting for the significant demographic or diagnostic covariates.
Mean Difference in PTGI pre- to post-session and pre- to post-intervention | through study completion, an average of 5 years
  The Post-Traumatic Growth Inventory (PTGI) examines the post-trauma growth using 21 items. The aim is to assess for statistically significant changes pre- to post session (1 day = a session) and pre- to post-intervention using paired t-test as well as ANCOVA adjusting for the significant demographic or diagnostic covariates.
Mean Difference in B-SCS pre- to post-session and pre- to post-intervention | through study completion, an average of 5 years
  The Brief Suicide Cognitions Scale (B-SCS) assesses the suicide risk. The aim is to assess for statistically significant changes pre- to post session (1 day = a session) and pre- to post-intervention using paired t-test as well as ANCOVA adjusting for the significant demographic or diagnostic covariates.

SECONDARY OUTCOMES:
Mean Difference in AAQII pre- to post-session | through study completion, an average of 5 years
  AAQII is a 10-item measure that assesses psychological flexibility, with higher values indicating greater psychological inflexibility. The aim is to assess for statistically significant changes between post sessions using the repeated measure ANOVA.
Mean Difference in PANAS pre- to post-session | through study completion, an average of 5 years
  PANAS measures short-term positive and negative emotions. The aim is to assess for statistically significant changes between post sessions using the repeated measure ANOVA.
Mean Difference in STAI pre- to post-session | through study completion, an average of 5 years
  The STAI tracks the symptoms of anxiety, and the total score ranges from 20 to 80. The aim is to assess for statistically significant changes between post sessions using the repeated measure ANOVA.

CONTACTS AND LOCATIONS:
Overall Officials: William Marchand, MD, Principal Investigator — VA Salt Lake City HCS
Locations (1):
- George E. Wahlen Department of Veterans Affairs Medical Center, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No